CLINICAL TRIAL: NCT03807869
Title: Efficacy and Safety of I-stent By-pass Implantation in Eyes With Open Angle Glaucoma
Brief Title: Reduction of Intraocular Pressure After I-stent By-pass Implantation in Eyes With Open Angle Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Bialystok (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1772
Record Dates: First submitted 2019-01-15; First posted 2019-01-17 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Glaucoma
Keywords: I-stent; glaucoma surgery; minimally invasive glaucoma surgery
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- coexisting glaucoma and cataract (Experimental): Patients with coexisting glaucoma and cataract qualified to combined glaucoma surgery
  Interventions: Procedure: combined glaucoma surgery

INTERVENTIONS:
Procedure: combined glaucoma surgery — phacoemulsification of cataract and I-stent by-pass implantation

SUMMARY:
Purpose of this study is to exam the hypotensive effectiveness of I-stent implantation depended on number of antiglaucoma eye drops at baseline.

DETAILED DESCRIPTION:
The scientific aim of the project is to estimate the average reduction of intraocular pressure (IOP) in relation to the initial number of antiglaucoma drops at the end of 12 months observation period. The subject must suffer from glaucoma and cataract at the same time, and qualify for a cataract surgery. The group will be composed of 40 patients of the Ophthalmology Clinic of the Medical University of Białystok qualified for planned cataract removal surgery. They will be surgically implanted an I-stent by-pass during phacoemulsification.

ELIGIBILITY:
Inclusion Criteria:

* co-existing glaucoma and cataract (NC1, NC2) classified by means of the LOCS III scale (Lens Opacity Classification System III)
* patients with primary open-angle glaucoma (POAG), pseudoexfoliative glaucoma (PGX) and normal tension glaucoma (NTG), with topical hypotensive treatment
* written consent to involvement and participation in the study for a period of at least 12 months was obtained from all patients after they had first been informed of the nature of the procedure and other surgical alternatives

Exclusion Criteria:

* no consent to participation in the study
* prior surgical and laser procedures in the area of the eye
* narrow- or closed-angle glaucoma
* post-inflammatory or post-traumatic secondary glaucoma
* chronic illness of the cornea or optic nerve
* advanced macular degeneration
* active inflammatory process
* pregnancy
* systemic steroid therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
IntraOcular Pressure measurement (IOP) | baseline, 12 months
  change in the level of intraocular pressure measured with Goldmann applanation tonometer
Best Corrected Visual Acuity measurement (BCVA) | baseline, 12 months
  change in best corrected visual acuity measured with Snellen charts

SECONDARY OUTCOMES:
number of antiglaucoma medicines | baseline, 12 months
  change in number of antiglaucoma medicines used before and after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Zofia Mariak, Prof, Study Chair — Medical University of Bialystok
Locations (1):
- Medical University, Bialystok, Poland

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months of study completion
Access Criteria: Data access requests will be reviewed by the Chair Person. Requestors will be required to sign a Data Access Agreement

REFERENCES:
- [Background] Myers JS, Masood I, Hornbeak DM, Belda JI, Auffarth G, Junemann A, Giamporcaro JE, Martinez-de-la-Casa JM, Ahmed IIK, Voskanyan L, Katz LJ. Prospective Evaluation of Two iStent(R) Trabecular Stents, One iStent Supra(R) Suprachoroidal Stent, and Postoperative Prostaglandin in Refractory Glaucoma: 4-year Outcomes. Adv Ther. 2018 Mar;35(3):395-407. doi: 10.1007/s12325-018-0666-4. Epub 2018 Feb 23. PMID 29476443
- [Result] Chansangpetch S, Lau K, Perez CI, Nguyen N, Porco TC, Lin SC. Efficacy of Cataract Surgery With Trabecular Microbypass Stent Implantation in Combined-Mechanism Angle Closure Glaucoma Patients. Am J Ophthalmol. 2018 Nov;195:191-198. doi: 10.1016/j.ajo.2018.08.003. Epub 2018 Aug 8. PMID 30098352
- [Derived] Kozera M, Konopinska J, Mariak Z, Rekas M. Effectiveness of iStent Trabecular Microbypass System Combined with Phacoemulsification versus Phacoemulsification Alone in Patients with Glaucoma and Cataract Depending on the Initial Intraocular Pressure. Ophthalmic Res. 2021;64(2):327-336. doi: 10.1159/000511456. Epub 2020 Sep 9. PMID 32906138
- [Derived] Konopinska J, Kozera M, Krasnicki P, Mariak Z, Rekas M. The Effectiveness of First-Generation iStent Microbypass Implantation Depends on Initial Intraocular Pressure: 24-Month Follow-Up-Prospective Clinical Trial. J Ophthalmol. 2020 Jun 23;2020:8164703. doi: 10.1155/2020/8164703. eCollection 2020. PMID 32676205